CLINICAL TRIAL: NCT00699556
Title: Do Treatments for Smoking Cessation Affect Alcohol Drinking? Study 1: Nicotine Replacement Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC0508000486; R01AA015596 (NIH)
Record Dates: First submitted 2007-12-25; First posted 2008-06-18 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Alcohol Drinking
Keywords: alcohol; nicotine; smoking cessation; smoking cessation medications
MeSH Terms: conditions — Alcohol Drinking; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patch+spray (Experimental): Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + nicotine nasal spray.
  Interventions: Drug: 21mg transdermal nicotine patch (Nicoderm CQ); Drug: 1mg nicotine nasal spray
- patch+placebo spray (Placebo Comparator): Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + placebo nicotine nasal spray.
  Interventions: Drug: 21mg transdermal nicotine patch (Nicoderm CQ); Drug: placebo nasal spray

INTERVENTIONS:
Drug: 21mg transdermal nicotine patch (Nicoderm CQ) — 21mg transdermal nicotine patch
  Other Names: Nicoderm CQ
Drug: 1mg nicotine nasal spray — two 0.5mg/sprays, one to each nostril (dose = 1mg) The nicotine nasal spray is formulated by the Investigational Drug Service at Yale-New Haven Hospital. It is similar in concentration to Nicotrol.
  Arms: patch+spray
Drug: placebo nasal spray — saline combined with capsaicin to mimic the brief nasal irritation from active nicotine spray The placebo nasal spray is formulated by the Investigational Drug Service at Yale-New Haven Hospital.
  Arms: patch+placebo spray

SUMMARY:
This study examines the effect of combined nicotine replacement therapy (transdermal patch + nasal spray vs. transdermal patch + placebo nasal spray) on reactivity to alcohol and self-administration behavior.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21 and over
* Able to read and write in English
* Smoker
* Heavy drinker

Exclusion Criteria:

* Any significant current medical or psychiatric conditions that would contraindicate the consumption of alcohol or nicotine
* Significant hepatocellular injury
* Positive test result at intake appointments on urine drug screens conducted for opiates, cocaine, or benzodiazepines
* Women who are pregnant or nursing
* Suicidal, homicidal, or evidence of severe mental illness
* Prescription of any psychotropic drug in the 30 days prior to study enrollment
* Blood donation within the past 8 weeks
* Individuals who are seeking treatment for drinking or smoking who have attempted to quit drinking or smoking within the past 3 months
* Specific exclusions for administration of nicotine nasal spray not specified above including nasal polyps, chronic nasal congestion, allergies, sinusitis
* Specific exclusions for administration of nicotine patch not specified above including history of dermatoses
* Reported sensitivity or allergies to pepper or pepper spray, peppermint, or prior adverse reaction to nicotine spray
* Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center & Yale-New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Patch+Spray First, Then Nicotine Patch+Placebo Spray; Nicotine Patch+Placebo Spray First, Then Nicotine Patch+Spray: Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + nicotine nasal spray and the other session they receive nicotine patch + placebo nasal spray. The order is counter-balanced.
  21mg transdermal nicotine patch (Nicoderm CQ): 21mg transdermal nicotine patch
  1mg nicotine nasal spray: two 0.5mg/sprays, one to each nostril (dose = 1mg)
  The nicotine nasal spray is formulated by the Investigational Drug Service (IDS) at Yale-New Haven Hospital. It is similar in concentration to Nicotrol.
  Or
  Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + placebo nicotine nasal spray.
  21mg transdermal nicotine patch (Nicoderm CQ): 21mg transdermal nicotine patch
  placebo nasal spray: saline combined with capsaicin to mimic the brief nasal irritation from active nicotine spray. Formulated by IDS at Yale.
Period: First Intervention (1 Day)
Arm/Group | Nicotine Patch+Spray First, Then Nicotine Patch+Placebo Spray | Nicotine Patch+Placebo Spray First, Then Nicotine Patch+Spray
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Nicotine Patch+Spray First, Then Nicotine Patch+Placebo Spray | Nicotine Patch+Placebo Spray First, Then Nicotine Patch+Spray
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Patch + Nicotine Spray; Nicotine Patch+Placebo Spray: Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + nicotine nasal spray and the other session they receive nicotine patch + placebo nasal spray. The order is counter-balanced.
  21mg transdermal nicotine patch (Nicoderm CQ): 21mg transdermal nicotine patch
  1mg nicotine nasal spray: two 0.5mg/sprays, one to each nostril (dose = 1mg)
  The nicotine nasal spray is formulated by the Investigational Drug Service (IDS) at Yale-New Haven Hospital. It is similar in concentration to Nicotrol.
  Or
  Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + placebo nicotine nasal spray.
  21mg transdermal nicotine patch (Nicoderm CQ): 21mg transdermal nicotine patch
  placebo nasal spray: saline combined with capsaicin to mimic the brief nasal irritation from active nicotine spray. Formulated by IDS at Yale.
Arm/Group | Nicotine Patch + Nicotine Spray; Nicotine Patch+Placebo Spray
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Consumed During an Ad-libitum Drinking Period
Description: Participants are presented with alcohol beverages and allowed to drink at their leisure.
Time Frame: Two hour ad-libitum drinking period during laboratory session
Measure: Mean (Standard Deviation); unit: drinks
Groups:
- Nicotine Patch+Nicotine Spray: Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + nicotine nasal spray.
  21mg transdermal nicotine patch (Nicoderm CQ): 21mg transdermal nicotine patch
  1mg nicotine nasal spray: two 0.5mg/sprays, one to each nostril (dose = 1mg) The nicotine nasal spray is formulated by the Investigational Drug Service at Yale-New Haven Hospital. It is similar in concentration to Nicotrol.
- Nicotine Patch+Placebo Spray: Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + placebo nicotine nasal spray.
  21mg transdermal nicotine patch (Nicoderm CQ): 21mg transdermal nicotine patch
  placebo nasal spray: saline combined with capsaicin to mimic the brief nasal irritation from active nicotine spray The placebo nasal spray is formulated by the Investigational Drug Service at Yale-New Haven Hospital.
Arm/Group | Nicotine Patch+Nicotine Spray | Nicotine Patch+Placebo Spray
Number analyzed (Participants) | 22 | 22
drinks | 1.59 (2.24) | 1.64 (2.30)

2. Secondary Outcome: Craving for Alcohol
Description: Alcohol craving was measured using the Alcohol Urge Questionnaire (AUQ). The range of scores is 1-100 on a visual analog scale (VAS). Higher scores indicate higher levels of craving. Score indicated is the total score.
Time Frame: first measurement during laboratory session (+60 minutes after beginning of laboratory session)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Nicotine Patch+ Nicotine Spray: Within subject design. All volunteers complete two laboratory sessions. In one session they receive nicotine patch + nicotine nasal spray.
  21mg transdermal nicotine patch (Nicoderm CQ): 21mg transdermal nicotine patch
  1mg nicotine nasal spray: two 0.5mg/sprays, one to each nostril (dose = 1mg) The nicotine nasal spray is formulated by the Investigational Drug Service at Yale-New Haven Hospital. It is similar in concentration to Nicotrol.
Arm/Group | Nicotine Patch+ Nicotine Spray | Nicotine Patch+Placebo Spray
Number analyzed (Participants) | 22 | 22
units on a scale | 14.75 (2.10) | 17.03 (2.33)

ADVERSE EVENTS:
Time Frame: During laboratory session, subjects responded to a list of potential symptoms. Symptoms were assessed 5 hours after nicotine administration.
Arm/Group | Patch+Spray | Patch+Placebo Spray
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 17/22 | 11/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patch+Spray (N=22) | Patch+Placebo Spray (N=22)
Skin Irritation (General disorders) | 1 | 0
Heart rate > 100 (Cardiac disorders) | 1 | 1
Dizziness/light headed (General disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 0 | 0
Abdominal discomfort (General disorders) | 1 | 0
Nasal irritation (General disorders) | 17 | 11
Throat irritation (General disorders) | 13 | 1
Eyes watering (General disorders) | 17 | 10
hands or feet cold (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No